CLINICAL TRIAL: NCT05191927
Title: A Nomogram Model to Predict Central Lymphnode Metastasis in Thyroid Papillary Carcinoma Suitable for Primary Hospitals
Brief Title: A Nomogram Model to Predict Central Lymphnode Metastasis in Thyroid Papillary Carcinoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Other Study IDs: NO.SYSEC-KY-KS-2021-180
Record Dates: First submitted 2021-11-17; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Thyroid Papillary Carcinoma
Keywords: Thyroid Papillary Carcinoma; nomogram; central lymph node metastasis; predictor
MeSH Terms: conditions — Thyroid Cancer, Papillary | interventions — Calcification, Physiologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- female group: all are female
- male group: all are male
  Interventions: Other: male

INTERVENTIONS:
Other: male — Nine preoperative predictors were identified for the nomogram: gender, age, platelet counts, TPOAb level and US signatures including maximum diameter, boundary, component, calcification and cervical lymph node enlargement.
  Other Names: young; high platelet count; low TPOAb level; larger maximum diameter; unclear boundary; solidity; calcification; cervical lymph node enlargement
  Groups: male group

SUMMARY:
To establish and validate a suitable and practical nomogram for primary hospitals to predict the risk of central lymph node metastasis (CLNM) among thyroid papillary carcinoma (PTC) patients based on clinical and ultrasound characteristics among Chinese population，1000 PTC patients were retrospectively reviewed who underwent bilateral thyroidectomy or lobectomy plus central lymph node dissection（CLND） between June 2014 and September 2019 in Sun Yat-sen Memorial Hospital (Guangzhou, South China), and then LASSO regression analysis was performed to screen out the possible predictors. Another 200 PTC patients from the First Affiliated Hospital of Zhengzhou University (Zhengzhou, North China) who underwent bilateral thyroidectomy or lobectomy plus CLND between March 2019 and November 2020 were enrolled to construct the nomogram. The area under the receiver operating characteristic (ROC) curves (AUC), calibration curves and decision curve analysis (DCA) were used to evaluate the nomogram.

DETAILED DESCRIPTION:
1000 Patients who underwent total thyroidectomy or lobectomy and were diagnosed as PTC by pathological examination between June 2014 and September 2019 in Sun Yat-sen Memorial Hospital (Guangzhou, South China) and 200 patients in the First Affiliated Hospital of Zhengzhou University (Zhengzhou, North China) from March 2019 to November 2020 were selected as the subjects to construct the nomogram. 1000 patients were randomized at 7:3 and divided into a training set and a verification set. Besides, 200 cases that met the inclusion and exclusion criteria above-mentioned in the First affiliated Hospital of Zhengzhou University were enrolled as a external verification set.

The following clinical features for each patient were obtained before surgery: gender, age, occupation, complicated with autoimmune diseases (absent / present), history of radiation exposure (absent / present), family history of thyroid cancer (absent / present), with other tumors (absent / present) and preoperative laboratory examinations including neutrophil count, lymphocyte count, platelet count, thyroid-stimulating hormone (TSH), free triiodothyronine (fT3), free thyroxine (fT4), anti-thyroglobulin antibody (TgAb), thyroid peroxidase antibody (TPOAb).

Preoperative US signatures of thyroid tumors were also included: distribution (unilateral / bilateral), shape (regular / irregular), maximum diameter, number (single / multiple), boundary（clear /heliclear / unclear), component (solid /cystic-solid), calcification (absent / microcalcification / macrocalcification), blood flow (absent / internal / annular), cervical lymph node enlargement (absent / present).

A nomogram were established for predicting CLNM based on the universally available baseline Characteristics of PTC patients at a tertiary hospital in South China and externally validate it with data from North China. Odd ratios (ORs), 95% confidence interval (CI) and probability values were obtained by logistic regression analysis. The area under the receiver operating characteristic (ROC) curve (AUC) was calculated to evaluate the accuracy of the nomogram for predicting CLNM. The calibration curve and Hosmer-Lemeshow tests were performed to evaluate the calibration of the nomogram. The decision curve analysis (DCA) was applied to validate clinical utility of the nomogram.

ELIGIBILITY:
Inclusion Criteria:

* underwent TC operation for the first time
* confirmed as PTC by postoperative pathological examination
* underwent ipsilateral or bilateral CLND

Exclusion Criteria:

* complicated with other subtypes of TC or thyroid metastatic cancer
* received preoperative interventional therapy (such as radiofrequency and microwave therapy) or head and neck radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent total thyroidectomy or lobectomy and were diagnosed as PTC by pathological examination in Sun Yat-sen Memorial Hospital (Guangzhou, South China) and in the First Affiliated Hospital of Zhengzhou University (Zhengzhou, North China) .
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Multivariate logistic regression analysis | 1day
  Multivariate logistic regression analysis were conducted to determine the potential nonlinear association between predictors and and the risk of CLNM.

CONTACTS AND LOCATIONS:
Overall Officials: mingtong xu, professor, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT05191927/Prot_SAP_000.pdf